CLINICAL TRIAL: NCT02411201
Title: DOTAREM® Pharmacokinetics, Safety and Efficacy Study in Pediatric Subjects Aged <2 Years (Term Newborn Infants to Toddlers 23 Months of Age Inclusive)
Brief Title: DOTAREM Pharmacokinetics and Safety Study in Pediatric Subjects Aged < 2 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DGD-44-063; 2013-003215-21 (EudraCT Number)
Record Dates: First submitted 2015-03-11; First posted 2015-04-08 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Magnetic Resonance Imaging
MeSH Terms: interventions — gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DOTAREM (Experimental)
  Interventions: Drug: DOTAREM

INTERVENTIONS:
Drug: DOTAREM — Single intravenous injection of 0.1 mmol/kg body weight
  Other Names: gadoterate meglumine

SUMMARY:
The main purpose of the study is to evaluate the pharmacokinetics of DOTAREM® in the body of children aged less than 2 years thanks to several blood samples (3 ml in total) taken following the administration of DOTAREM®.

DOTAREM® is a contrast agent commonly used for enhancement of Magnetic Resonance Imaging (MRI) to potentially improve the quality of the images and help the diagnosis. Children aged less than 2 years scheduled to undergo routine gadolinium-enhanced MRI of any body region may take part in the study. In this case they will receive DOTAREM®, a solution injected at the standard dose of 0.2mL/kg (0.1 mmol/kg) of body weight.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subject aged <2 years (term newborn infants to toddlers 23 months of age inclusive). Term is defined as ≥37 weeks of amenorrhea
* Subject is scheduled to undergo routine gadolinium-enhanced MRI of any body region (e.g. CNS, cardiac) at the dose of 0.1 mmol/kg BW (0.2 mL/kg BW)
* Subject with normal renal function for its age, estimated glomerular filtration rate calculated based on the Schwartz formula

Exclusion Criteria:

* Subject planned for intervention (e.g. surgery) between the screening visit and up to 24 hours after DOTAREM injection
* Subject whose preceding or subsequent treatment to DOTAREM injection (e.g., blood loss or receiving blood, treatment with diuretics, etc…) would alter DOTAREM pharmacokinetics parameters
* Subject with subsequent planned treatment after DOTAREM injection that would prevent obtaining the required blood samples (e.g., emergency surgery, etc…)
* Subject with a history of a bleeding disorder
* Subject with severe liver disease (Child's Pugh Classification B or greater or serum direct bilirubin greater than 0.3 mg/dL, age adjusted)
* Subject with electrolyte or fluid imbalance that presents undue risk
* Subject undergoing a change in chemotherapy within 48 hours prior to and up to 24 hours after DOTAREM injection
* Subject who received or will receive any other contrast agent within 72 hours prior to DOTAREM injection or up to 24 hours after DOTAREM injection
* Subject with contraindication for MRI such as iron metal implants (e.g. aneurysm clips)
* Subject with history of anaphylactoid or anaphylactic reaction to any allergen including drugs and contrast agents
* Subject having participated within 30 days in a clinical study involving an investigational drug or device
* Subject planned to participate simultaneously to another clinical study

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Project Manager, Study Director — Guerbet
Locations (9):
- Landes-Frauen-und Kinderklinik Linz, Linz, Austria
- France (3):
  - CHU, Bordeaux
  - CHRU, Lille
  - Hôpital de Hautepierre, Strasbourg
- Hungary (3):
  - Department of Molecular and Neurological Clinical and Research Center, Budapest
  - University of Debrecen Medical Center, Debrecen
  - Borsod-Abaúj-Zemplén University County Hospital, Miskolc
- Poland (2):
  - Uniwersytecki Szpital Dziecięcy w Lublinie, Lublin
  - Instytut Pomnik -Centrum Zdrowia Dziecka, Warsaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 children aged less than 2 years were recruited in 4 countries: Austria, France, Hungary and Poland.
Groups:
- DOTAREM: Subjects receiving a single intravenous injection of 0.1 mmol/kg body weight of DOTAREM
Period: Overall Study
Arm/Group | DOTAREM
Started | 51
Completed | 45
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Age group completed | 2

BASELINE CHARACTERISTICS:
Population: 51 pediatric subjects were included in the study. 4 subjects could not be randomized due to consent withdrawal (n=1), adverse event (n=1) or other reason (n=2). 2 subjects did not receive DOTAREM due to consent withdrawal for 1 subject and adverse event for the second subject.
Arm/Group | DOTAREM
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: months] | 9.9 (7.4)
Age, Customized [Count of Participants; unit: Participants]
  <1 month | 5
  1 to 3 months | 9
  >3 months to <24 months | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 22
Region of Enrollment [Number; unit: participants]
  Austria | 3
  Hungary | 9
  Poland | 29
  France | 4

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of DOTAREM in Plasma
Description: Pharmacokinetics interpretation was performed using a pharmacokinetic population modelling approach. DOTAREM concentrations in plasma were analyzed using a validated LC-MS/MS method. Area under the curve was determined from typical and individual DOTAREM concentration-time profiles.
Time Frame: Blood samples were collected during 3 time windows: 15 min to 60 min, 2 hours to 4 hours and 6 hours to 8 hours post-injection
Population: Among the 45 subjects who received one injection of DOTAREM, all had at least one blood sample available for pharmacokinetics.
Measure: Median (Full Range); unit: hour.µmol/L
Arm/Group | DOTAREM
Number analyzed (Participants) | 45
hour.µmol/L | 1591.1 [981.43 to 2841]

2. Primary Outcome: Rate Constant of the Terminal Phase of DOTAREM
Description: Pharmacokinetics interpretation was performed using a pharmacokinetic population modelling approach. DOTAREM concentrations in plasma were analyzed using a validated LC-MS/MS method. Rate constant of the terminal phase was determined from typical and individual DOTAREM concentration-time profiles.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour-1
Arm/Group | DOTAREM
Number analyzed (Participants) | 45
hour-1 | 0.5117 [0.2288 to 0.7824]

3. Primary Outcome: Terminal Elimination Half-life of DOTAREM From Plasma
Description: Pharmacokinetics interpretation was performed using a pharmacokinetic population modelling approach. DOTAREM concentrations in plasma were analyzed using a validated LC-MS/MS method. Terminal elimination half-life was determined from typical and individual DOTAREM concentration-time profiles.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: hour
Arm/Group | DOTAREM
Number analyzed (Participants) | 45
hour | 1.3545 [0.8859 to 3.0291]

4. Primary Outcome: Total Clearance of DOTAREM From Plasma
Description: Pharmacokinetics interpretation was performed using a pharmacokinetic population modelling approach. DOTAREM concentrations in plasma were analyzed using a validated LC-MS/MS method. Total clearance was determined from typical and individual DOTAREM concentration-time profiles.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: L/hour per kg
Arm/Group | DOTAREM
Number analyzed (Participants) | 45
L/hour per kg | 0.0602 [0.0352 to 0.1019]

5. Primary Outcome: Volume of Distribution of DOTAREM at Steady State
Description: Pharmacokinetics interpretation was performed using a pharmacokinetic population modelling approach. DOTAREM concentrations in plasma were analyzed using a validated LC-MS/MS method. Volume of distribution at steady state was determined from typical and individual DOTAREM concentration-time profiles.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: L/kg
Arm/Group | DOTAREM
Number analyzed (Participants) | 45
L/kg | 0.0473 [0.0273 to 0.1597]

6. Secondary Outcome: Simulated Plasma Concentration of DOTAREM
Description: Pharmacokinetics interpretation was performed using a pharmacokinetic population modelling approach. DOTAREM concentrations in plasma were analyzed using a validated LC-MS/MS method.
Time Frame: at 10 and 20 min post-injection
Population: as for outcome 1
Measure: Median (Full Range); unit: µmol/L
Arm/Group | DOTAREM
Number analyzed (Participants) | 45
µmol/L
  Simulated concentration at 10 min | 320.92 [45.223 to 2857]
  Simulated concentration at 20 min | 275.67 [47.048 to 1565.1]

7. Secondary Outcome: MRI Lesion Visualization at Subject Level
Description: Lesion visualization was assessed on up to five most representative lesions per subject based on scoring of 3 co-endpoints:
  * border delineation (based on a 3-point scale where 1=none; 2=moderate and 3=clear and complete)
  * internal morphology (based on a 3-point scale where 1=poorly visible; 2=moderately visible and 3=sufficiently visible)
  * contrast enhancement (based on a 3-point scale where 1=none; 2=weak and 3=clear and bright)
  For each co-endpoint, a sum of scores was calculated at subject level as follows: sum of scores = score of the lesion 1 (+ score of the lesion 2 + score of the lesion 3 + score of the lesion 4 + score of the lesion 5, when applicable)
Time Frame: Pre-injection and post-injection (estimated between 5 and 20 minutes after injection)
Population: Lesion visualization was evaluated in 28 subjects who underwent contrast-enhanced MRI for central nervous system indication.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pre-contrast: Lesion visualization was assessed before DOTAREM injection
- Pre- + Post-contrast: Lesion visualization was assessed after DOTAREM injection
Arm/Group | Pre-contrast | Pre- + Post-contrast
Number analyzed (Participants) | 28 | 28
units on a scale
  Sum of scores of lesion border delineation | 4.3 (3.7) | 5.1 (4.0)
  Sum of scores of internal morphology | 4.3 (3.9) | 5.2 (4.3)
  Sum of scores of contrast enhancement | 1.9 (1.5) | 5.0 (4.5)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from informed consent signature to the end of the study (7+/-1 day after DOTAREM administration)
Arm/Group | DOTAREM
Serious Adverse Events (participants affected / at risk) | 1/45
Other Adverse Events (participants affected / at risk) | 12/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOTAREM (N=45)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOTAREM (N=45)
Pyrexia (General disorders) | 5 (5)
Device difficult to use (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All written or oral papers and publications must have the joint agreement of the investigator and Guerbet.

The Investigator shall not use the sponsor's name in any publication without the prior permission of Guerbet.

Each investigator agrees not to publish/present the evaluation of the main criterion involving only the patients he/she has included.

Any abstract project will be first submitted to Guerbet at least 10 working days before submission to the congress scientific committee.